CLINICAL TRIAL: NCT06144151
Title: A Pilot Study for Pupillary Assessment to Predict CAR-T Related Neurotoxicity
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0176; NCI-2023-09804 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Neurotoxicity
MeSH Terms: conditions — Neurotoxicity Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: NeurOptics® NPi®-300 Pupillometer — The pupilometer is a non-invasive device which will be placed in front of your eyes, one at a time. It looks like a handheld spotlight or scanner, with a small plastic guide sticking out that will be placed against your cheek to help keep the device in place during the scan. It will not touch your eye. Both your left and right eyes will be measured with the device each time. Scanning with the pupilometer will take less than 5 minutes total for both eyes.

SUMMARY:
To learn about the relationship between changes in pupil size and reactivity and the start of neurological side effects in patients after receiving CAR-T cell therapy.

DETAILED DESCRIPTION:
Primary Objective:

To assess the association between the status of NPi drop from baseline (prior to CAR T-cell infusion) to the lowest NPi post Axi-cel (CD19 CAR-T cell) infusion and the status of immune effector cell-associated neurotoxicity onset within 10 days post CD19 CAR-T cell infusion.

Secondary Objective:

To evaluate the largest absolute difference in NPi between two eyes (∆ NPi) and assess its association with severity of clinical symptoms as measured by Immune Effector Cell Encephalopathy (ICE) and or radiographic / EEG findings

Exploratory Objective:

To assess the feasibility and safety of a pupillometer use in patient treated with Axi-cel therapy.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for study participation, patient will satisfy all relevant inclusion criteria and none of the exclusion criteria.

Inclusion Criteria:

1. Ages Eligible for Study: 18 Years and above (Adult, Older Adult)
2. Sexes Eligible for Study: All
3. Patient with histologically proven DLBCL, PMBCL or tFL, or follicular Lymphoma receiving axi-cel CAR-T cell therapy in the inpatient setting at MD Anderson Cancer Center
4. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have already been administered CAR-T cell therapy.
2. The patient who is unwilling or unable to comply with the requirements of the study including being able to be assessed with pupillometer
3. Patient has a condition which places him at an unacceptable risk as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Ranjit Nair, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org